CLINICAL TRIAL: NCT00913588
Title: Comparative, Randomized, Single-Dose, 3-way Crossover Bioavailability Study of Geneva and Dista (Prozac) 20 mg Fluoxetine Hydrochloride Capsules (Pulvules) In Health Adult Males Under Fed and Fasted Conditions Following Administration of a 40 mg Dose
Brief Title: To Demonstrate the Relative Bioavailability of Geneva and Dista (Prozac) 20 mg Fluoxetine Hydrochloride Capsules (Pulvules) In Healthy Adult Males Under Fed and Fasted Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Eric Mittleberg, Ph.D, VP of Product Development, Sandoz Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 960379
Record Dates: First submitted 2009-06-02; First posted 2009-06-04 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2009-06

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Fluoxetine

ARMS (3):
- 1 (Experimental): Fluoxetine HCl 20 mg Capsules Under Fasting Conditions (Geneva Pharmaceutical, Inc.)
  Interventions: Drug: Fluoxetine HCl 20 mg Capsules Under Fasting Conditions (Geneva Pharmaceutical, Inc.)
- 2 (Experimental): Fluoxetine HCl 20 mg Capsules Under Fed Conditions (Geneva Pharmaceutical, Inc.)
  Interventions: Drug: Fluoxetine HCl 20 mg Capsules Under Fed Conditions (Geneva Pharmaceutical, Inc.)
- 3 (Active Comparator): Prozac Fluoxetine HCl 20 mg Capsules Under Fed Conditions (Dista)
  Interventions: Drug: Prozac Fluoxetine HCl 20 mg Capsules Under Fed Conditions (Dista)

INTERVENTIONS:
Drug: Fluoxetine HCl 20 mg Capsules Under Fasting Conditions (Geneva Pharmaceutical, Inc.)
  Arms: 1
Drug: Fluoxetine HCl 20 mg Capsules Under Fed Conditions (Geneva Pharmaceutical, Inc.)
  Arms: 2
Drug: Prozac Fluoxetine HCl 20 mg Capsules Under Fed Conditions (Dista)
  Arms: 3

SUMMARY:
To demonstrate the relative bioavailability of Geneva and Dista (Prozac) 20 mg Fluoxetine Hydrochloride capsules (Pulvules) in healthy adult males under fed and fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal finding on physical exam, medical history, or clinical laboratory results on screening.

Exclusion Criteria:

* Positive test results for HIV or hepatitis B or C.
* Treatment for drug or alcohol dependence.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 1996-05; Primary Completion 1996-08 (Actual); Study Completion 1996-08 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on AUC and Cmax | 141 days

CONTACTS AND LOCATIONS:
Overall Officials: Roderick Malone, M.D., Principal Investigator — Clinical Research Center (Cincinnati)